CLINICAL TRIAL: NCT00707629
Title: Long Term Effects of Diabetes of Very Young Children
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Principal Investigator, Linda DiMeglio, MD, MD, Indiana University
Other Study IDs: 0507-18
Record Dates: First submitted 2008-06-30; First posted 2008-07-01 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes; neurocognitive measures; behavioral measures
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Insulin Pump Therapy: Children on insulin pumps for at least three years. Subjects must have type 1 diabetes for at least five years and diagnosed under the age of 5.

SUMMARY:
To investigate neurocognitive and behavioral measures in 25 children aged 6-10 years diagnosed with diabetes for > 5 years who have received long-term insulin pump therapy (> 3 years) compared to a group of children matched for age, sex, glycemic control, and diabetes duration treated with insulin injections. Outcome measures will assess: clinical variables, cognitive status (intelligence, neuropsychological functioning), academic achievement, behavior, parenting stress, and quality of life.

It is hypothesized that long term insulin pump therapy initiated during early childhood can delay the progression of neurocognitive complications of diabetes, decrease parental stress, and improve school performance and quality of life, as compared to insulin injections.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have type 1 diabetes for at least 5 years, diagnosed prior to the age of 5 years
* Children recruited on pumps must have used pump therapy for at least 3 years
* Parents/guardians must be understand the protocol and be able to give consent, with assent obtained from all children over the age of 7 years.

Exclusion Criteria:

* Children will be excluded if they have additional medical problems requiring treatment with agents known to affect blood glucose such as steroids or L-asparaginase.
* Children must not have any other chronic illness in addition to diabetes with the exception of treated autoimmune hypothyroidism.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children between ages 6 and 10. Diagnosed with type 1 diabetes prior to the age of 5 years.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2005-08; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Diabetes Control | Data Collected at each study visit
  HbA1c, number of severe low events, frequency of moderate and mild hypoglycemia, blood glucose averages, and variance of reported blood sugar
Ease of Injections versus Insulin pump Therapy | Conclusion of study
  Mechanical issues, site infections and errors of insulin administration

CONTACTS AND LOCATIONS:
Overall Officials: Linda A DiMeglio, MD, Principal Investigator — Indiana University/Riley Hospital for Children
Locations (1):
- Riley Hospital for Children, Indianapolis, Indiana, United States